CLINICAL TRIAL: NCT01880502
Title: A Randomized, Double-blind, Placebo-controlled, Single-dose, Dose Escalation Study (Phase I) to Evaluate the Tolerability and Pharmacokinetics of Belviq in Adult Korean Volunteers
Brief Title: Pharmacokinetic Study of Belviq in Adult Korean Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: IlDong Pharmaceutical Co Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: ID_Belviq_1301
Record Dates: First submitted 2013-06-12; First posted 2013-06-19 (Estimated); Last update posted 2013-10-14 (Estimated); Status verified 2013-10

CONDITIONS: Healthy
Keywords: Healthy, Volunteers
MeSH Terms: interventions — lorcaserin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Belviq 10mg (Experimental)
  Interventions: Drug: Belviq 10mg
- Belviq 20mg (Experimental)
  Interventions: Drug: Belviq 20mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Belviq 10mg — Belviq 10mg single dose administration
  Arms: Belviq 10mg
Drug: Belviq 20mg — Belviq 20mg single dose administration
  Arms: Belviq 20mg
Drug: Placebo — Placebo single dose administration
  Arms: Placebo

SUMMARY:
A randomized, double-blind, placebo-controlled, single-dose, dose escalation study (Phase I) to evaluate the tolerability and pharmacokinetics of Belviq in adult Korean volunteers.

DETAILED DESCRIPTION:
The volunteers are screened through medical history, physical exam, laboratory tests etc. within 4 weeks (-28d~-2d) prior to the day scheduled for taking the investigational product (1d). The final subjects determined eligible for this clinical trial through screening tests are randomized to the dose groups with Belviq 10 mg and 20 mg. Twelve subjects are assigned to each group (9 subjects to study drug and 3 subjects to placebo), and the study drug or placebo are administered to the corresponding administration group. The subjects are discharged on the morning of 4d after completing the set study schedule at 72 hours after administration. The subjects then visit for the final tests on the last out-patient visiting day. Belviq is progressed sequentially from the low-dose group to the high-dose group.

The blood sampling time for the pharmacokinetic evaluation is as follows. Blood sampling for pharmacokinetic evaluation

: Before administration(0), and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 16, 24, 36, 48 and 72 h (17 times) after medication.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a healthy adult aged 18 ~ 60 years old at the time of screening.
2. Subject has body weight index (BMI) 23.0 ~ 32.0.

   ☞ BMI(kg/m2) = weight (kg)/{height (m)}2
3. Subject does not have congenital or chronic disease and is without pathologic symptom or finding on medical exam.

   Vital sign Supine SBP (mmHg) 90-140 DBP (mmHg) 50-90 Heart rate (beat/min) 40-80 Respiratory rate (breaths/min) 8-18
4. Subject was determined eligible according to the results of clinical laboratory tests like serum test, hematologic test, blood chemistry test, urine test etc. and vital signs, electrocardiography, physical exam etc. performed during the screening exam.

   SBP(mmHg) 90-140 DBP(mmHg) 50-90 Heart rate (beat/min) 40-80 Respiratory rate (breaths/min) 8-18
5. Subject decided to participate voluntarily and gave written Informed consent to comply with the instructions after listening to and fully understanding the detailed explanation about this trial.

Exclusion Criteria:

1. Subject has clinically significant liver, kidney, neurologic, immunologic, respiratory, endocrine disease or hematologic·oncologic disease, cardiovascular disease or psychiatric disease (mood disorder, compulsive disorder etc.) or such medical history (including subject with hepatitis virus in case of liver disease).
2. Subject has history of gastrointestinal disease (such as Crohn's disease, ulcer, acute or chronic pancreatitis etc.) or gastrointestinal surgery (except simple appendectomy or hernia operation) that can affect the absorption of the study drug.
3. Subject has hypersensitivity reaction to drug (aspirin, antibiotics etc.) or history of clinically significant hypersensitivity reaction.
4. Subject has history of drug abuse or tested positive to abused drug in the urine drug screening test (performed during screening and on Day -1).
5. Subject took any prescribed drug or oriental medicine within 2 weeks prior to the first medication or any over-the-counter (OTC) drug or vitamins within 1 week prior to the first medication or paracetamol 48 hours prior to taking the study drug (however, the subject can be included if other criteria are met according to the discretion of the investigator).
6. Subject participated in another study and received medication within 3 months prior to the first medication day (3 months are judged to be the period in between medications).
7. Subject has history of using the following drug

   * Fenfluramine/dexfenfluramine or phentermine
   * Drug that may increase the risk of valvulopathy or primary pulmonary hypertension (Cyproheptadine, Trazodone, Nefazodone, Amoxapine, tricyclic antidepressants, mirtazapine, pergolide, ergotamine, methysergide).
8. Subject received whole blood transfusion (500 mL) within 3 months prior to the first medication or blood transfusion within 1 month prior to the first medication.
9. Subject continually drinks (in excess of 28 units/week (21 unit/week for women), 1 unit = 10 g of pure alcohol) or cannot abstain from drinking for 48 hours prior to the study drug administration through the hospitalization period.
10. Subject smokes 3 cigarettes or more in one day or cannot abstain from smoking for 48 hours prior to the study drug administration through the hospitalization period.
11. Subject took caffeine-containing food within 48 hours prior to the first medication, or cannot abstain from taking during the hospitalization period.
12. Subject has tested positive to HbsAg, HCV Ab, HIV Ab tests.
13. Subject has peculiar diet, is a vegetarian or consumes food that may affect the drug metabolism (e.g. St. John's Wort).
14. Subject had serious change in dietary habit or activity from 4 weeks prior to the study drug administration.
15. Subject or his/her partner cannot or is not willing to use appropriate contraceptives during the trial period and for 28 days after termination of the study (for women, exclusion criteria include pregnant or breastfeeding woman or woman who was confirmed to be pregnant in the pregnancy test).
16. Subject was judged not to be eligible according to the discretion of the investigator for other reasons.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2013-06; Primary Completion 2013-07 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Vital signs | participants will be followed for the duration of hospital stay and post study visit, an expected average of 10 days
adverse event | participants will be followed for the duration of hospital stay and post study visit, an expected average of 10 days
electrocardiography | participants will be followed for the duration of hospital stay and post study visit, an expected average of 10 days
clinical laboratory tests | participants will be followed for the duration of hospital stay and post study visit, an expected average of 10 days
physical exam | participants will be followed for the duration of hospital stay and post study visit, an expected average of 10 day
echocardiography | participants will be followed for the duration of hospital stay and post study visit, an expected average of 10 days

SECONDARY OUTCOMES:
Change in Belviq concentration in the blood with time | Before administration(0), and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 16, 24, 36, 48 and 72 h (17 times) after medication.
Cmax, Cmax/D, AUClast, AUClast/D, AUCinf, AUCinf/D, tmax, t1/2 of Belviq | Before administration(0), and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 16, 24, 36, 48 and 72 h (17 times) after medication.
CL/F, Vz/F of Belviq | Before administration(0), and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 16, 24, 36, 48 and 72 h (17 times) after medication

CONTACTS AND LOCATIONS:
Overall Officials: Kyoung Sang You, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Jongno-gu, Seoul, South Korea